CLINICAL TRIAL: NCT03660969
Title: Heart&Muscle Study
Brief Title: Reliability of Cardiac Troponins for the Diagnosis of Myocardial Infarction in the Presence of Skeletal Muscle Disease
Acronym: H&M
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Cantonal Hospital of Aarau, Switzerland (Other); Medical University Innsbruck (Other); University Hospital, Zürich (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: BASEL XII; Research Grant (Other Grant/Funding Number: Swiss Heart Foundation)
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Myopathy; Muscle Weakness; Muscle Damage; Muscle Spasticity; Muscle Cramp; Muscle Injury; Muscle Soreness; Muscle Atrophy
Keywords: troponin
MeSH Terms: conditions — Muscular Diseases; Muscle Weakness; Muscle Spasticity; Muscle Cramp; Myalgia; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, muscle biopsies when clinically available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Visits to the emergency department (ED) for chest pain are extremely common and require a safe, rapid and efficacious treatment algorithm to exclude a possible AMI. These diagnostic algorithms are partly based on an important laboratory value, which showed growing utility in the diagnostic and prognostic of many cardiovascular diseases in the last years : cardiac troponin.

However, some patients with muscle disease often present with unexplained elevated high-sensitive cardiac Troponin T (hs-cTnT) levels in the absence of cardiac disease. The investigators aim at the characterization of the behaviour of this biomarker and its alternative (high-sensitive cardiac Troponin I), which will have important clinical implications on patients management.

DETAILED DESCRIPTION:
Introduction: The detection of cardiomyocyte injury as quantified by blood concentrations of cardiac troponin T (cTnT) or I (cTnI) is central in the diagnosis of acute myocardial infarction (AMI). While multiple cardiac disorders other than AMI may also lead to cardiomyocyte injury and therefore elevations in cTnT and cTnI, latest generations of cTnT and cTnI assays are considered to have near exclusive cardiac-specificity. Overall, both analytes (cTnT and cTnI) seem to have comparable diagnostic accuracy among patients presenting with suspected AMI to the emergency department (ED). However, their use in the diagnosis of AMI in patients with a skeletal muscle disease is questioned, as especially cTnT was found to be elevated in this setting. These increased cTnT levels have been successively attributed to a possible re-expression of cTnT isoforms in the diseased muscle, to a primary cardiac involvement associated with the muscle disease or to a cross-reaction of the hs-cTnT assay with TnT of muscle origin.

Aim: To characterize cTn levels in patients with a skeletal muscle disease to assess their utility in the field of cardiology (through their implication in AMI diagnosis and their diagnostic and prognostic accuracy regarding a possible cardiac involvement) and in the field of neurology (for the detection and risk-stratification of the muscle disorder itself).

Methodology: This study will be conducted at the University Hospital of Basel, at the Kantonsspital Aarau, both in Switzerland, and at the University Hospital of Innsbruck, Austria. A prospective cohort patient will be recruited through the neurology, rheumatology and cardiology clinics of these three hospitals. This prospective cohort of patients presenting with skeletal muscle disease will allow us to systematically screen patients for cTn increases, to investigate the prevalence and characteristics of a possible primary cardiac involvement (as documented by electrocardiogram, echocardiography, magnetic resonance imaging, cTnI, NT-proBNP (N-terminal pro-B-type Natriuretic Peptide) and any available further cardiac testing) and to explore the origins of the elevated cTn levels using muscle biopsies. Furthermore, this prospective cohort will document the role of these biomarkers in the diagnosis, prognosis and risk-stratification of the muscle disease. Patients will receive a 1- and 3-year follow-up visit with blood draw in order to measure cTn and other biomarkers and record the impact of the evolution and treatment of the muscle disease on these levels. Major adverse cardiac events including cardiovascular death, AMI, hospitalization for heart failure, and the development of clinical or subclinical heart failure as quantified by elevated blood concentrations of NT-proBNP will be recorded during follow-up.

Potential significance: Elevated cTnT levels do not only have consequences regarding the diagnosis of AMI but also raise many questions regarding their possible use as a diagnostic, prognostic and risk-stratification marker regarding the different muscle injuries and their possible primary cardiac involvement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic or suspicion of muscle disease as presence of specified keyword in patient's file or as screened by colleagues of the rheumatology, neuromuscular or other medical clinics.
* Patient consent available

Exclusion Criteria:

* Patient's refusal
* Age <18 years old
* Terminal kidney insufficiency with need for dialysis.
* Temporary exclusion criteria : Acute health condition such as myocardial infarction, patients presenting with a major trauma, a sepsis, patients shortly after cardiac surgery, and patients in shock (>100 bpm, <90 systolic BP, evidence of organ dysfunction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive participants which have been or currently are in treatment for a muscle disease at the University hospital of Basel, at the Canton Hospital of Aarau, University Hospital of Zürich or Bern or at the Medical University of Innsbruck, or who received a new diagnosis/suspicion of such a disease will be included.
Sampling Method: Probability Sample
Enrollment: 797 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of cTnT and cTnI levels as measured by different hs-cTn assays in patients with skeletal muscle disease. | 1 year

SECONDARY OUTCOMES:
Comparison of levels of cTnT and cTnI as measured by hs-assays in matched patients with and without skeletal muscle disease. | 1 year
Regression model of diverse patients' characteristics on levels of hs-cTnI and hs-cTnT in the context of skeletal muscle disease versus no skeletal muscle disease. | 1 year
Prognostic value of hs-cTn levels in patients with and without skeletal muscle disease. | 3 years
Characterization of cTnT and cTnI on skeletal muscle biopsies from myopathic patients. | 1 year
Characterization of the impact of cTnT and cTnI on the diagnosis and prognosis of muscle diseases | 3 years
  Prognosis defined as the incidence of Major Cardiovascular Events (MACE is defined as a composite of death, acute myocardial infarction, life-threatening arrhythmia (cardiac arrest, sustained ventricular tachycardia, atrioventricular (AV) -block III), cardiac arrest/reanimation, acute heart failure (requiring admission to a hospital or intra-hospital transfer to the intensive care unit), stroke/transient ischemic attack, pulmonary embolism)

OTHER OUTCOMES:
Research on the development of a new cTnT-assay | 3 years
Protein characterization | 3 years
Cardiac troponin as predictors or screening tools for a cardiac involvement | 3 years
Cardiac troponin as predictor of evolution and therapeutic response of the muscle disease or muscle regeneration. | 3 years
Characterisation of cardiac troponin in diseases of various etiologies involving muscles | 3 years
Impact of muscle symptoms on cardiac troponin | 3 years
Cardiac troponin versus other markers (e.g. CK) of inflammation/necrosis of peripheral muscles. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mueller, MD, Principal Investigator — University Hospital, Basel, Switzerland; Angelika Hammerer, MD, Principal Investigator — Canton Hospital Aarau; Julia Wanschitz, MD, Principal Investigator — Medical University Innsbruck
Locations (5):
- Medical University Innsbruck, Innsbruck, Austria
- Switzerland (4):
  - Canton Hospital of Aarau, Aarau, Canton of Aargau
  - University Hospital Basel, Basel
  - Inselspital Bern, Bern
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schmid J, Liesinger L, Birner-Gruenberger R, Stojakovic T, Scharnagl H, Dieplinger B, Asslaber M, Radl R, Beer M, Polacin M, Mair J, Szolar D, Berghold A, Quasthoff S, Binder JS, Rainer PP. Elevated Cardiac Troponin T in Patients With Skeletal Myopathies. J Am Coll Cardiol. 2018 Apr 10;71(14):1540-1549. doi: 10.1016/j.jacc.2018.01.070. PMID 29622161
- [Background] Jaffe AS, Vasile VC, Milone M, Saenger AK, Olson KN, Apple FS. Diseased skeletal muscle: a noncardiac source of increased circulating concentrations of cardiac troponin T. J Am Coll Cardiol. 2011 Oct 18;58(17):1819-24. doi: 10.1016/j.jacc.2011.08.026. Epub 2011 Sep 29. PMID 21962825
- [Derived] du Fay de Lavallaz J, Prepoudis A, Wendebourg MJ, Kesenheimer E, Kyburz D, Daikeler T, Haaf P, Wanschitz J, Loscher WN, Schreiner B, Katan M, Jung HH, Maurer B, Hammerer-Lercher A, Mayr A, Gualandro DM, Acket A, Puelacher C, Boeddinghaus J, Nestelberger T, Lopez-Ayala P, Glarner N, Shrestha S, Manka R, Gawinecka J, Piscuoglio S, Gallon J, Wiedemann S, Sinnreich M, Mueller C; BASEL XII Investigators. Skeletal Muscle Disorders: A Noncardiac Source of Cardiac Troponin T. Circulation. 2022 Jun 14;145(24):1764-1779. doi: 10.1161/CIRCULATIONAHA.121.058489. Epub 2022 Apr 7. PMID 35389756